CLINICAL TRIAL: NCT01567475
Title: A Phase I/II Study Investigating the Combination of RAD001 and Rituximab in Patients With Non-Hodgkin's Lymphomas
Brief Title: The Combination of Rad001 and Rituximab In Patients With Non-hodgkin's Lymphomas
Acronym: (RAD001-R)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD001-R
Record Dates: First submitted 2011-10-26; First posted 2012-03-30 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Non-Hodgkin's Lymphomas
MeSH Terms: interventions — Everolimus; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus and rituximab (Experimental)
  Interventions: Drug: Everolimus and rituximab

INTERVENTIONS:
Drug: Everolimus and rituximab — One injection of Rituximab 375 mg/m2 per week during 28 days followed by one Rituximab infusion every other cycle at 375 mg/m2 associated with everolimus at 5mg or 10 mg every day or 5 mg every other day.

SUMMARY:
This study is an open label, multicenter study with two phases:

* Phase I is a dose escalation study of RAD001 in combination with one injection of Rituximab 375 mg/m² per week during 4 weeks (28 days) in patients CD20 positive non-Hodgkin's lymphomas to determine the dose limiting toxicities (DLTs) and maximum tolerated dose (MTD). The purpose of the study is to assess the feasibility of the combination based on - rate of dose limiting toxicities (DLT) and PK drug-drug interaction (DDI).
* Phase II will define the efficacy and safety profile of RAD001 and Rituximab combination at the RP2D in patients with lymphomas.

Patients with lymphomas will be treated at the RP2D established during phase I and evaluated for clinical benefit rate, comprising complete responses (CR + CRu), partial responses (PR) and stable disease (SD), and time to progression using the IWG criteria for treatment response.

Induction therapy will follow the same schedule than during the phase I study.

Maintenance therapy: Monthly cycles for up to 2 years with:

* Daily RAD001 at the same dose than during induction therapy.
* Rituximab infusion every other cycle at 375 mg/m2 that correspond to the usual maintenance schedule for Rituximab.

Response to therapy will be assessed between day 42 and day 49, then every two months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory of one of the following CD 20 positive B-cell Lymphoma:

  * Mantle cell, Marginal zone, lymphocytic, follicular lymphoma
  * Histological transformation from low grade to high grade
* Must have had at least one previous chemotherapy regimen and not more than 5 previous chemotherapy regimens.
* Disease is measurable: existence of a bidimensional lesion greater than 2 cm in its longer diameter or malignant lymphocytosis greater than 5000 x 109/L
* Recovery from any non-hematological toxicity derived from previous treatments. The presence of alopecia and NCI-CTC grade < 2 symptomatic peripheral neuropathy is allowed.
* Age ≥18 years old;
* Eastern Co-operative Oncology Group (ECOG) performance status 0-1;
* Adequate liver and renal function, defined by total bilirubin ≤2.5 x institutional upper limit of normal (ULN) or ≤5 x ULN if liver is involved by malignancy as judged by the investigator (explanation must be provided) and creatinine ≤ 221 μmol/L ;
* Fasting serum cholesterol ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Adequate bone marrow function, defined by absolute neutrophil count (ANC) ≥1000/mm3 and platelet count ≥100,000/mm3, unless due to disease;
* At least 3 weeks since previous chemotherapy, biological therapy, radiation therapy, major surgery, or other investigational cancer therapy that is considered disease-directed and have recovered from prior toxicities to Grade 0-1;
* All men of reproductive potential and women† of child-bearing potential (WOCBP) must agree to practice effective contraception during the entire study period and for one month after the last study treatment, unless documentation of infertility exists.

  † A woman patient is considered to have childbearing potential unless she meets at least one of the following criteria 1) Age > 50 years and naturally amenorrhoeic for > 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential); or 2) Premature ovarian failure confirmed by a specialist gynaecologist or 3) Previous bilateral salpingo-oophorectomy, or hysterectomy, or 4) XY genotype, turner syndrome, uterine agenesis.
* Able to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* Uncontrolled clinically significant inter-current illness including, but not limited to, ongoing to active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients receiving antibiotics for infections that are under control may be included in the study;
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients receiving chronic, systemic treatment with corticosteroids (at a dose equivalent or greater than 20 mg prednisone per day) or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * symptomatic congestive heart failure of New York heart Association Class III or IV
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy.)
  * active (acute or chronic) or uncontrolled severe infections
  * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
* Leptomeningeal or uncontrolled CNS localization
* Concurrent malignancy, except patients with early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, localized prostate cancer, or cervical intraepithelial neoplasia;
* Treatment with any other investigational drugs within the preceding 4 weeks
* Known HIV-positive (since such patients are at increased risk of lethal infections when treated with potentially marrow-suppressive therapy);
* Known active hepatitis A, B, or C, or history of hepatitis A, B or C;
* Women who are pregnant or lactating
* Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to everolimus or other rapamycin (e.g., sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimen
* Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Phase I part: Determination of the Recommended Dose of RAD001 in combination with rituximab. | 28 days
  Determination of recommended dose will be based on safety parameters and particularly on incidence of DLTs .
Phase II part: Complete Response Rate (CR+CRu) | 2 years
  Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma Cheson,1999)

SECONDARY OUTCOMES:
OVERALL RESPONSE RATE | 2 years
  The same disease response assessment used for complete response rate will be considered to determine the Overall Response Rate. Patient is defined as a responder if he/she has a complete response (CR/CRu) or partial response (PR) at the end of treatment. A descriptive analysis will also be performed considering as nonresponders all patients who relapsed or died during treatment phase even if they were prematurely withdrawn as responder.
PROGRESSION-FREE SURVIVAL | Up to 4 years
  Progression-Free Survival will be measured from the date of inclusion to the date of first documented disease progression, relapse or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.
OVERALL SURVIVAL | Up to 4 years
  Overall survival will be measured from the date of inclusion to the date of death from any cause. Patients who are alive at the time of analysis will be censored at the date of the last contact.
DURATION OF RESPONSE | Up to 4 years
  Duration of response will be measured from the date of first documentation of a response (CR/CRu or PR after induction or at the end of treatment) to the date of first documented evidence of progression/relapse or death from any cause. Responding patients and patients who are lost to follow up will be censored at their last tumor assessment date.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIBRAG, Doctor, Principal Investigator — Service Hématologie, Institut Gustave Roussy
Locations (5):
- France (5):
  - Service des Maladies du Sang - CHRU de Lille, Lille
  - Service Hématologie - Hôtel Dieu de NANTES, Nantes
  - Service Hématologie - CHU Lyon Sud, Pierre-Bénite
  - Service Hématologie - Centre Henri Becquerel, Rouen
  - Service Hématologie - Institut Gustave Roussy, Villejuif

REFERENCES:
- See also: LYSA Lymphoma : The LYmphoma Study Association — http://www.lysa-lymphoma.org/